CLINICAL TRIAL: NCT01190358
Title: Grape Seed Extract and Postprandial Oxidation and Inflammation: A Pilot Study in People With the Metabolic Syndrome.
Brief Title: Grape Seed Extract and Postprandial Oxidation and Inflammation
Acronym: GSEMetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 200917488
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Grape Seed Extract; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Dietary Supplement: Placebo
- Grape seed extract (Active Comparator): 300mg of grape seed extract.
  Interventions: Dietary Supplement: Grape seed extract

INTERVENTIONS:
Dietary Supplement: Placebo — Sugar pill containing maltodextrin.
  Other Names: Placebo, non-active components
  Arms: Placebo
Dietary Supplement: Grape seed extract — Meganatural Gold® contains 300mg of grape seed extract.
  Other Names: Active, Meganatural Gold®
  Arms: Grape seed extract

SUMMARY:
The purpose of this study is to determine whether taking grape seed extract prior to eating a high fat meal will reduce the inflammatory response in people with the metabolic syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether taking grape seed extract prior to eating a high fat meal will reduce the inflammatory response in people with the metabolic syndrome. If this extract is shown to mitigate the inflammatory response induced by a high fat meal, it could potentially aid in postponing of the diagnosis of diabetes or other chronic diseases associated with high levels of inflammation.

ELIGIBILITY:
Inclusion Criteria:

The metabolic syndrome will be diagnosed on the basis of having a combination of any 3 of the following factors:

1. Waist circumference of ≥ 40 inches (men) or ≥ 35 inches (women)
2. Elevated triglycerides ≥150mg/dl
3. HDL cholesterol of < 40mg/dl (men) or < 50mg/dl (women)
4. Elevated blood pressure of ≥ 130/85mmHg
5. Fasting glucose of > 100mg/dL

Exclusion criteria:

* Smokers
* Female subjects who are pregnant or lactating
* Subjects taking any medications that would interfere with outcomes of the study i.e. lipid lowering medications, anti-inflammatory drugs (i.e. ibuprofen), dietary supplements
* Subjects with any known allergy or intolerance to foods involved in the study (cantaloupe, egg, dairy, wheat, grape seed extract)
* Subjects who are actively trying to lose weight
* Subjects with unusual dietary habits (i.e. pica, anorexia nervosa, extreme food restriction, binging and/or purging disorders)
* Subjects who are addicted to drugs or alcohol or who are <1 year recovery program
* Subjects who present with significant psychiatric or neurological disturbances as determined by the primary investigator (i.e. uncontrolled bipolar disorder)
* Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, uncontrolled hypertension (≥ 140/90mmHg), liver and kidney disease as identified by routine blood tests (chemistry panels). These subjects will be referred to their primary care doctor for further care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Modification of the postprandial inflammatory response. | 7 hours
  Analysis of inflammatory markers known to increase following a meal high in fat (~40% kcal from fat). Markers to be analyzed will include the following:
  1. Serum lipids
  2. Oxidized LDL
  3. Hs-CRP
  4. TNFα
  5. IL1
  6. IL6

SECONDARY OUTCOMES:
Metabolic response to a high fat meal. | 7 hours
  Assay for the insulin and glucose response generated from consumming a high fat meal (~40% of kcal from fat).

CONTACTS AND LOCATIONS:
Overall Officials: Chulani T Kappagoda, M.D., Ph. D., Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis (Academic Surge, Ragle Human Nutrition Research Facility), Davis, California
  - VA Hospital, Mather, Mather, California